CLINICAL TRIAL: NCT01443936
Title: Phase 1 Study of Safety and Immunogenicity of Ad4-H5-VTN in Ad4 Seronegative and Seropositive Volunteers
Brief Title: Experimental AD4-H5-VTN Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110259; 11-I-0259
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-04-24

CONDITIONS: H5N1 Influenza
Keywords: Influenza Vaccine; H5N1 Influenza; Normal Volunteer; Adenovirus; Live Virus Vaccine; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza, Human; Adenoviridae Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: Ad4-H5-VTN vaccination-tonsillar route
Biological: Ad4-H5-vaccination-oral route

SUMMARY:
This is a Phase 1 randomized, single center, dose-escalation study designed to evaluate the safety and immunogenicity of live, replication competent recombinant Adenovirus type 4-H5N1Influenza Vietnam 1194 Hemagglutinin (HA) (Ad4-H5-Vtn). Determining the optimal route and dose for this recombinant platform will greatly accelerate investigations of this vector as an influenza vaccine and an HIV vaccine platform.

Intranasal and tonsillar administration of the vaccine will be separately assessed. The oral enteric-coated capsule will also be assessed in 10 outpatients using similar blood sampling for comparison. The Ad4-H5-Vtn orally administered as enteric-coated capsules has already been evaluated in an ascending dose Phase 1 study, in dosages as high as 10(11) viral particles (vp).

The primary goal of this study is to evaluate safety of ascending dosages of the Ad4-H5-Vtn vaccine following intranasal and tonsillar administration. A dosage or dosages will be selected to further evaluate the humoral, cellular, and mucosal immune responses against both the vector and the inserted gene. The Ad4-H5-Vtn will be initiated at 10(3) vp. Once safety is established at the initial dose, a second round of testing will begin at the next ten-fold higher dose. The Ad4-H5-Vtn vaccine will be assessed in three participants at each dosage level. The maximum viral dose administered by the tonsillar route will be 10(8) vp.

In addition to clinical and laboratory monitoring of safety, the principal assessments will be shedding of the Ad4-H5-Vtn virus in rectal, cervicovaginal, throat, and nasal swabs, and assessment of the antibody (mucosal and systemic) response to the HA and to the Ad4 virus. When safety has been confirmed in all three participants at a given dosage level, the next higher dose group is enrolled. If one grade 3 or greater toxicity (or pre-specified Grade 2 toxicity, see Section 3.4) attributable to the vaccine is observed, the group will be expanded at that dose. If a second attributable grade 3 or greater toxicity (or pre-specified Grade 2 toxicity, see Section 3.4) is observed, the dose will be reduced one level and the group will be expanded. Up to 25 Ad4-seronegative individuals will be enrolled at the maximum tolerated dose to fully evaluate safety and immunogenicity in the protocol.

All participants will be followed for 28 days following immunization, and again at 8 and 26 weeks to evaluate any long-term toxicity and persistence of immunity. Tonsillar Participants will receive a booster dose of vaccine [SK1]at the 26-week visit and be seen for follow-up visits at Weeks 30 and 34. Household and intimate contacts will also be enrolled and monitored for Adenovirus and HAI antibodies.

DETAILED DESCRIPTION:
This is a Phase 1 randomized, single center, dose-escalation study designed to evaluate the safety and immunogenicity of live, replication competent recombinant Adenovirus type 4-H5N1Influenza Vietnam 1194 Hemagglutinin (HA) (Ad4-H5-Vtn). Determining the optimal route and dose for this recombinant platform will greatly accelerate investigations of this vector as an influenza vaccine and an HIV vaccine platform.

Tonsillar administration of the vaccine will be separately assessed. The oral enteric-coated capsule will also be assessed in 10 outpatients using similar blood sampling for comparison. The Ad4-H5-Vtn orally administered as enteric-coated capsules has already been evaluated in an ascending dose Phase 1 study, in dosages as high as 10(11) viral particles (vp).

The primary goal of this study is to evaluate safety of ascending dosages of the Ad4-H5-Vtn vaccine following intranasal and tonsillar administration. A dosage or dosages will be selected to further evaluate the humoral, cellular, and mucosal immune responses against both the vector and the inserted gene. The Ad4-H5-Vtn will be initiated at 10(3) vp. Once safety is established at the initial dose, a second round of testing will begin at the next ten-fold higher dose. The Ad4-H5-Vtn vaccine will be assessed in three participants at each dosage level. The maximum viral dose administered by the tonsillar route will be 10(8) vp.

In addition to clinical and laboratory monitoring of safety, the principal assessments will be shedding of the Ad4-H5-Vtn virus in rectal, cervicovaginal, throat, and nasal swabs, and assessment of the antibody (mucosal and systemic) response to the HA and to the Ad4 virus. When safety has been confirmed in all three participants at a given dosage level, the next higher dose group is enrolled. If one grade 3 or greater toxicity (or pre-specified Grade 2 toxicity, see Section 3.4) attributable to the vaccine is observed, the group will be expanded at that dose. If a second attributable grade 3 or greater toxicity (or pre-specified Grade 2 toxicity, see Section 3.4) is observed, the dose will be reduced one level and the group will be expanded. Up to 25 Ad4-seronegative individuals will be enrolled at the maximum tolerated dose to fully evaluate safety and immunogenicity in the protocol.

All participants will be followed for 28 days following immunization, and again at 8 and 26 weeks to evaluate any long-term toxicity and persistence of immunity. All subjects will be offered to receive a booster vaccination with a recombinant hemagglutinin influenza H5 vaccine after the 26-week visit and be seen for follow-up visits 4 and 8 weeks following booster immunization, with an additional telephone follow-up 6 months after boosting. Household and intimate contacts will also be enrolled and monitored for Adenovirus and HAI antibodies following Ad4-H5-Vtn administration only; household and intimate contacts will not be enrolled or monitored during the boost portion of the study.

We will conduct an expansion H5N1 boost phase of this study, in which all vaccinees from the initial phase of the study will be offered re-enrollment to receive a booster vaccination with an FDA-approved H5N1 inactivated monovalent influenza vaccine. We will offer enrollment in the expansion phase to all participants who received the Ad4-H5-Vtn vaccine in the initial phase, regardless of whether they also received the recombinant hemagglutinin influenza H5 vaccine boost. We will also enroll individuals who have never received an H5 influenza vaccine as controls. Participants will receive a single vaccination with the H5N1 vaccine and be seen for follow-up visits 4 and 8 weeks later for immunogenicity evaluations.

ELIGIBILITY:
* INCLUSION CRITERIA

All participants (vaccinees, household contacts, and intimate contacts) must meet all of the following criteria:

1. Age 18 to 49 years for vaccinees. Vaccinees may be >49 years of age at the time of booster vaccination. Age 18 to 65 years for household and intimate contacts.
2. Negative FDA-approved HIV test
3. Able to provide proof of identity to the acceptance of the Principal Investigator or designee during enrollment.
4. Available and willing to participate in follow-up visits and tests for the duration of the study,
5. Willing to have samples stored for future research.
6. Negative <=-HCG pregnancy test for females presumed to be of reproductive potential.
7. A female must meet one of the following criteria:

   1. No reproductive potential because of menopause (one year without menses) or because of a

      hysterectomy, bilateral oophorectomy, or tubal ligation.

      or
   2. Participant agrees to be heterosexually inactive or consistently practice contraception at least 21 days

   prior to enrollment and 28 days following vaccination. Acceptable methods of contraception

   include the following:
   * condoms, male or female, with a spermicide
   * diaphragm or cervical cap with spermicide
   * contraceptive pills, Norplant, or Depo-Provera
   * male partner has previously undergone a vasectomy for which there is documentation.
   * intrauterine device
8. Male participants must agree to practice abstinence or effective birth control for at least 21 days prior to enrollment and during the first 28 days following vaccination.

The following inclusion criteria apply only to vaccinees and not to household or intimate contacts:

1. Willing to receive HIV test results and abide by NIH guidelines for partner notification of positive HIV results.
2. Physical examination and laboratory results without clinically significant findings within the 8 weeks prior to enrollment.
3. Willing to avoid vaccination other than the study agent for 30 days prior to and 30 days after administration of the Ad4-H5-Vtn vaccine.
4. Safety Laboratory Criteria within 8 weeks prior to enrollment:

   * Hematopoietic: White blood cell count and Lymphocyte count +/- 25% the normal limits for the NIH Clinical Center
   * Platelet count of least 125,000/mm3
   * Hemoglobin >11.2 g/dL for females and >13.0 g/dL for males.
   * Renal: BUN <23 mg/dL; creatinine within normal limits for the NIH Clinical Center
   * Hepatic: Serum total bilirubin 2 mg/dL
   * Metabolic: ALT <2 times upper limit of normal range
   * Endocrine: Serum glucose within normal range
5. Additional Laboratory Criteria:

   * Immunologic: No history of hypogammaglobulinemia
   * Serologic: Ad4 neutralizing antibody 80% inhibitory dilution <1:100

The following inclusion criteria apply only to tonsillar vaccinees and not to oral vaccine recipients,

household contacts, or intimate contacts:

1. Either no history of tonsillectomy OR the presence of tonsils on physical exam.

INCLUSION CRITERIA FOR THE EXPANSION H5N1 BOOST PHASE:

1. Age 18 to 64.
2. Negative pregnancy test (women of childbearing potential).
3. Group-specific inclusion criteria:

   * For participants in the study group: prior receipt of the Ad4-H5-Vtn vaccine in the initial phase of this study.
   * For participants in the control group: no prior receipt of an H5 vaccine product (by self-report).

EXCLUSION CRITERIA

A participant (vaccinees, household contacts, and intimate contacts) will be excluded if they have the following:

1. Any condition that, in the investigator's judgement, places the subject at undue risk by participating in the study.

The following exclusion criterion applies to vaccinees and intimate contacts, but not to household contacts:

1. History of any prior disease or therapy which would affect immune or pulmonary function.
2. Prior malignancy, except curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
3. History of radiation therapy or cytotoxic/cancer chemotherapy.
4. History of insulin-dependent diabetes mellitus.
5. Immunodeficiency or autoimmune disease.
6. Acute infection or a recent (within 6 months) history of chronic infection suggestive of immunodeficiency.
7. Taking any medication which may affect immune function, except participants may be taking low doses of nonprescription strength NSAIDS (including e.g. ibuprofen or aspirin) or acetaminophen.
8. Chronic respiratory disorders including asthma, emphysema, interstitial lung disease, pulmonary hypertension, recurrent pneumonia, or recent or ongoing respiratory tract infection. If a respiratory disorder is transient, defer immunization but do not exclude the participant.
9. Active Hepatitis B or C infection, as indicated by the presence of Hepatitis B antigen or Hepatitis C virus (i.e. Hepatitis B or C positive serology with the presence of virus antigen or DNA. Ongoing viral

   replication will be confirmed by a Hepatitis B antigen or Hepatitis C viral load).
10. Female of child-bearing potential who is breast-feeding or planning pregnancy during the 28 days following vaccination.

The following exclusion criteria apply only to vaccinees and not to household or intimate contacts:

1. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to receipt of live virus vaccine, protocol adherence, or a participant s ability to give informed consent.
2. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.
3. Participants that live in the same house or apartment with any of the following will be excluded:

   * An individual under 18 years of age
   * An immunocompromised or immunosuppressed individual
   * An individual with chronic respiratory disease
   * A woman who is currently pregnant or planning a pregnancy during the period of immunization
4. Healthcare worker who has direct contact with immunodeficient, unstable patients, or pediatric patients.
5. Participants caring for children <36 months of age. Potential vaccinees with any household or intimate contact who cares for children <36 months of age will also be excluded.
6. Receipt of any of the following:

   * Antiviral medications within 30 days prior to vaccination
   * Blood products within 120 days prior to HIV screening
   * Immunoglobulin within 60 days prior to HIV screening
   * Investigational research drugs or any other investigational agent that in the judgement of the PI might interact with the study vaccine within 30 days prior to initial study vaccine administration
   * Allergy treatment with antigen injections within 30 days of study vaccine administration
7. History of Guillain-Barr(SqrRoot)(Copyright) syndrome.
8. History of H5 influenza vaccination.

EXCLUSION CRITERIA FOR THE EXPANSION H5N1 BOOST PHASE:

1. History of systemic hypersensitivity reactions to egg proteins or life-threatening reactions to previous influenza vaccinations.
2. History of Guillain-Barr(SqrRoot)(Copyright) syndrome.
3. Acute infection or a recent (within 6 months) history of chronic infection suggestive of immunodeficiency.
4. Taking any medication which may affect immune function, except participants may be taking low doses of nonprescription strength NSAIDS (including e.g. ibuprofen or aspirin) or acetaminophen.
5. Receipt of an approved vaccine, investigational research drugs, or any other investigational agent that in the judgement of the PI might interact with the study vaccine within 30 days prior to H5N1 vaccine administration.
6. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to receipt of the H5N1 vaccine, protocol adherence, or a participant s ability to give informed consent.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-09-14; Primary Completion 2018-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Safety: evaluate local toxicity & systemic reactions to vaccination. Severe reactions to vaccine (i.e. lower respiratory or GI tract disease) or systemic symptoms related to vaccine.

SECONDARY OUTCOMES:
Immunogenicity: Data collected for: H5-specific antibody, mucosal humoral, & cellular immune response; vaccine virus shedding & genetic stability; transmission of virus to household/intimate contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Connors, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Amara RR, Villinger F, Altman JD, Lydy SL, O'Neil SP, Staprans SI, Montefiori DC, Xu Y, Herndon JG, Wyatt LS, Candido MA, Kozyr NL, Earl PL, Smith JM, Ma HL, Grimm BD, Hulsey ML, Miller J, McClure HM, McNicholl JM, Moss B, Robinson HL. Control of a mucosal challenge and prevention of AIDS by a multiprotein DNA/MVA vaccine. Science. 2001 Apr 6;292(5514):69-74. doi: 10.1126/science.1058915. PMID 11393868
- [Background] Baba TW, Jeong YS, Pennick D, Bronson R, Greene MF, Ruprecht RM. Pathogenicity of live, attenuated SIV after mucosal infection of neonatal macaques. Science. 1995 Mar 24;267(5205):1820-5. doi: 10.1126/science.7892606.
- [Background] Baba TW, Liska V, Khimani AH, Ray NB, Dailey PJ, Penninck D, Bronson R, Greene MF, McClure HM, Martin LN, Ruprecht RM. Live attenuated, multiply deleted simian immunodeficiency virus causes AIDS in infant and adult macaques. Nat Med. 1999 Feb;5(2):194-203. doi: 10.1038/5557. PMID 9930868
- [Derived] Matsuda K, Migueles SA, Huang J, Bolkhovitinov L, Stuccio S, Griesman T, Pullano AA, Kang BH, Ishida E, Zimmerman M, Kashyap N, Martins KM, Stadlbauer D, Pederson J, Patamawenu A, Wright N, Shofner T, Evans S, Liang CJ, Candia J, Biancotto A, Fantoni G, Poole A, Smith J, Alexander J, Gurwith M, Krammer F, Connors M. A replication-competent adenovirus-vectored influenza vaccine induces durable systemic and mucosal immunity. J Clin Invest. 2021 Mar 1;131(5):e140794. doi: 10.1172/JCI140794. PMID 33529172